CLINICAL TRIAL: NCT05359068
Title: A Multi-center, Randomized, Double-blind, Double-Dummy, Positive Parallel Controlled Study to Evaluate the Efficacy and Safety in Treatment of Mild-moderate Essential Hypertension
Brief Title: Study to Evaluate the Efficacy and Safety of SPH3127 In Patients With Mild-moderate Essential Hypertension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shanghai Pharmaceuticals Holding Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SPH3127-301
Record Dates: First submitted 2022-04-27; First posted 2022-05-03 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2023-06

CONDITIONS: Essential Hypertension
MeSH Terms: conditions — Essential Hypertension | interventions — SPH3127; Valsartan

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- Stage 1 Arm A (Experimental): 1 SPH3127 tablet，3 SPH3127 matching placebo tablets, 1 valsartan matching placebo capsule, once daily for 12 weeks.
  Interventions: Drug: SPH3127 tablet
- Stage 1 Arm B (Experimental): 2 SPH3127 tablets，2 SPH3127 matching placebo tablets, 1 valsartan matching placebo capsule, once daily for 12 weeks.
  Interventions: Drug: SPH3127 tablet
- Stage 1 Arm C (Experimental): 4 SPH3127 tablets, 1 valsartan matching placebo capsule, once daily for 12 weeks.
  Interventions: Drug: SPH3127 tablet
- Stage 1 Arm D (Experimental): 4 SPH3127 matching placebo tablets, 1 valsartan capsule, once daily for 12 weeks.
  Interventions: Drug: Valsartan
- Stage 2 Arm A (Experimental): 2 SPH3127 tablets, 1 valsartan matching placebo capsule, once daily for 12 weeks.
  Interventions: Drug: SPH3127 tablet
- Stage 2 Arm B (Experimental): 2 SPH3127 matching placebo tablets, 1 valsartan capsule, once daily for 12 weeks.
  Interventions: Drug: Valsartan
- Stage 3 (Experimental): 2 SPH3127 tablets, once daily for 40 weeks.
  Interventions: Drug: SPH3127 tablet

INTERVENTIONS:
Drug: SPH3127 tablet — 1 tablet
  Arms: Stage 1 Arm A
Drug: SPH3127 tablet — 2 tablets
  Arms: Stage 1 Arm B
Drug: SPH3127 tablet — 4 tablets
  Arms: Stage 1 Arm C
Drug: Valsartan — 1 valsartan capsule
  Arms: Stage 1 Arm D
Drug: SPH3127 tablet — 2 tablets
  Arms: Stage 2 Arm A; Stage 3
Drug: Valsartan — 1 valsartan capsule
  Arms: Stage 2 Arm B

SUMMARY:
The primary aim of the study is to assess the antihypertensive efficacy of SPH3127 in patients with mild to moderate essential hypertension.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female of age ≥18 years;
2. Diagnosed with mild-moderate essential hypertension;
3. Participant has understood the study-required procedures, voluntarily signed informed consent.

Exclusion Criteria:

1. Diagnosed with secondary hypertension, suspected grade 3 hypertension, acute hypertension, or at risk when current antihypertensive therapy discontinued;
2. Suffered by severe heart disease within 6 months;
3. Suffered by severe cerebrovascular disease within 6 months;
4. Suffered by severe or malignant retinopathy;
5. Out of controlled diabetes;
6. History of malignant tumor;
7. History of mental disorder;
8. Subject is planning or in use of other antihypertensive drugs or other drugs may affect blood pressure during the trial;
9. Alcohol or drug abuse;
10. Pregnant, lactating women or subject is planning to pregnant within 6 months after the trial;
11. Assessed by the investigators as unsuitable for participating in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 957 (Actual)
Dates: Start 2021-06-10 (Actual); Primary Completion 2023-12-26 (Actual); Study Completion 2023-12-26 (Actual)

PRIMARY OUTCOMES:
Change from baseline in mean sitting diastolic blood pressure (msDBP) at week 12 | Measure at week 12 of treatment.

SECONDARY OUTCOMES:
Changes from baseline in mean sitting diastolic blood pressure (msDBP) at week 2, 4, 6, 8 and 10 | Measured at week 2, 4, 6, 8 and 10 of treatment.
Changes from baseline in mean sitting diastolic blood pressure (msSBP) at week 2, 4, 6, 8, 10 and 12. | Measured at week 2, 4, 6, 8, 10, and 12 of treatment.
Total effective rate at week 2, 4, 6, 8, 10 and 12 | Measured at week 2, 4, 6, 8, 10, and 12 of treatment.
Rate of reaching target blood pressure at week 2, 4, 6, 8, 10 and 12 | Measured at week 2, 4, 6, 8, 10, and 12 of treatment.
Number of subjects with adverse event. | 12 weeks.
Plasma concentration of SPH3127. | 12 weeks.
Relationship between SPH3127 exposure and renin inhibition level/efficacy/adverse events | 12 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Changsheng Ma, Principal Investigator — Beijing Anzhen Hospital, Capitcal Medical University
Locations (40):
- China (40):
  - Beijing Hospital, Beijing, Beijing Municipality
  - Beijing Anzhen Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Beijing Pinggu Hospital, Beijing, Beijing Municipality
  - Affiliated Hospital of Chongqing Three Gorges Medical College, Chongqing, Chongqing Municipality
  - Lanzhou University Second Hospital, Lanzhou, Gansu
  - Guangdong Second Provincial General Hospital, Guangzhou, Guangdong
  - Guangdong Provincial People's Hospital, Guangzhou, Guangdong
  - Liuzhou people's Hospital, Liuchow, Guangxi
  - Hainan Third People's Hospital, Sanya, Hainan
  - Cangzhou Central Hospital, Cangzhou, Hebei
  - The First Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - The Third Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Luoyang Third People's Hospital, Luoyang, Henan
  - Henan Provincial People's Hospital, Zhengzhou, Henan
  - Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Tongji hospital,Tongji Medical college of HUST, Wuhan, Hubei
  - The Third Xiangya Hospital of Central South University, Changsha, Hunan
  - XiangYa Hospital CentralSouth University, Changsha, Hunan
  - The Second Xiangya Hospital of Central South University, Changsha, Hunan
  - The First Affiliated Hospital of Baotou Medical College, Inner Mongolia University of Science and Technology, Baotou, Inner Mongolia
  - Chifeng Municipal Hospital, Chifeng, Inner Mongolia
  - The Affiliated Hospital of Inner Mongolia Medical University, Hohhot, Inner Mongolia
  - The Second Affiliated Hospital of Nanjing Medical University, Nanjin, Jiangsu
  - The First Affiliated Hospital with Nanjing Medical University, Nanjing, Jiangsu
  - Suzhou Municipal Hospital, Suzhou, Jiangsu
  - The Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu
  - Xuzhou Central Hospital, Xuzhou, Jiangsu
  - Affiliated Hospital of Jiangsu University, Zhenjiang, Jiangsu
  - Shengjing Hospital of China Medical University, Shenyang, Liaoning
  - The People's Hospital of Liaoning Province, Shenyang, Liaoning
  - General Hospital of Ningxia Medical University, Yinchuan, Ningxia
  - The First People's Hospital of Yinchuan, Yinchuan, Ningxia
  - Ruijin Hospital, Shanghai Jiaotong University School Of Medicine, Shanghai, Shanghai Municipality
  - Yuncheng Central Hospital, Yuncheng, Shanxi
  - West China Hospital,Sichuan University, Chengdu, Sichuan
  - People's Hospital of Tianjin, Tianjin, Tianjin Municipality
  - Tianjin Fourth Central Hospital, Tianjin, Tianjin Municipality
  - The First Affiliated Hospital of Xinjiang Medical University, Ürümqi, Xinjiang
  - Affiliated Hangzhou First People's Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Zhejiang Provincial people's Hospital, Hangzhou, Zhejiang